CLINICAL TRIAL: NCT02890706
Title: Iodine Mapping Using Subtraction in Pulmonary Embolism Computed Tomography Versus Dual Energy Computed Tomography
Brief Title: Iodine Mapping Using Subtraction in Pulmonary Embolism CT Versus Dual-Energy CT
Acronym: InSPECT-DECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL56542.091.16
Record Dates: First submitted 2016-07-12; First posted 2016-09-07 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism (PE); Dual-Energy CT (DECT); Subtraction imaging
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Other): Each patient undergo the same CT protocol. Theobservers will observe the detection of the perfusion defects in two different techniques.
  Interventions: Device: Iodine Mapping using Subtraction in Pulmonary Embolism Computed Tomography versus Dual Energy Computed Tomography

INTERVENTIONS:
Device: Iodine Mapping using Subtraction in Pulmonary Embolism Computed Tomography versus Dual Energy Computed Tomography — Compare two techniques of the CT scanner

SUMMARY:
Comparing two techniques (Subtraction and Dual Energy CT) for functional Chest CT for patients with suspected with pulmonary embolism.

DETAILED DESCRIPTION:
Rationale: Iodine mapping of the lung using subtraction imaging in addition to standard computed tomography pulmonary angiography (CTPA) may improve the evaluation of pulmonary embolism (PE) in the same manner as the addition of dual energy computed tomography (DECT) to CTPA.

Objective: To evaluate image quality and accuracy of detection of perfusion defects associated with pulmonary pathology on iodine maps of the lung that are created by two different CT techniques: 1. A standard of care CTPA with DECT and 2. A new technique that subtracts a low radiation dose unenhanced CT from mono-energetic CTPA (subtraction) Study design: A maximum of 375 patients will undergo a standard CTPA with DECT according to local clinical guidelines, to have 30 patients with pulmonary embolism. For the purposes of this study, patients will undergo an additional unenhanced, low-radiation dose chest CT. Standard reconstructions of all scans and DECT iodine maps will be obtained for clinical reporting and subsequent treatment decisions, according to standard clinical routine. For research purposes, selected mono-energetic images will be post-processed using a novel subtraction algorithm to create iodine maps of the lungs. The iodine maps based on the subtraction algorithm will not be used for clinical management, only the additional unenhanced scan will be used in clinical management.

Study population: Patients presenting with a clinical indication for pulmonary CT angiography because of suspected pulmonary embolism. Only adult patients (≥ 35 years) who are able to provide informed consent will be enrolled.

Main study parameters/endpoints:

Main endpoint of the study is presence of perfusion as established by an expert panel with access to all imaging information (including CTPA, subtraction and DECT) and clinical follow-up. Accuracy of DECT and subtraction is established by observers who are blinded to CTPA and clinical data. Presence of iodine density differences in perfusion defects is measured using region of interest (ROI) measurements.

Images will be evaluated for objective and subjective image quality. Patient characteristics, radiation dose, clinical diagnosis, treatment decisions and patient outcome (all cause - and PE related mortality) will be recorded.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

CT imaging is associated with risks related to the use of radiation and iodinated contrast administration. No additional contrast will be used as compared to standard clinical practice as patients will only undergo one CTPA scan. The CT protocol of this study has been carefully designed to have a radiation dose identical or even lower than standard CT protocols for pulmonary embolism detection. The estimated dose-length product (DLP) of standard CTPA with DECT in Meander Medical Centre is 167 mGy-cm (effective dose is 2.4 mSv, using 0,0146 mSv/mGy-cm as a conversion factor). The researchers will expose patients who participate in the study to an estimated additional DLP of 72 mGy-cm due to the unenhanced scan, resulting in an additional estimated effective dose of 1,0 mSv. This implies that the total radiation dose is within the same range as radiation doses of other scans for PE detection in the Netherlands. The additional scan is not obligatory in pulmonary embolism diagnosis, but will be used for clinical evaluation of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients 35 years or older and able to provide informed consent
* Clinically requested CTPA because of suspected pulmonary embolism
* Available history and physical examination.

Exclusion Criteria:

* Pregnancy
* Hemodynamic instability
* Uncooperative patients.
* Contra-indication to intravenous iodine administration.
* Inability to position the arms above the shoulders

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Presence of perfusion defects as reference standard | 1.5 year
  After 1.5 year, the radiologists scores the presence of perfusion defects caused by pulmonary embolism as a reference standard.

SECONDARY OUTCOMES:
Radiation dose | Through study completion, an average of 2 months
Clinical diagnosis of Pulmonary embolism: after 6 months follow-up | Through study completion, after the first inclusion, the patients are followed for half a year.
30-day all cause mortality and PE-associated mortality | Through study completion, an average of three months
6 months all cause mortality and PE-associated mortality | Through study completion, an average of three months

CONTACTS AND LOCATIONS:
Overall Officials: Monique Brink, MD, Study Chair — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deak PD, Smal Y, Kalender WA. Multisection CT protocols: sex- and age-specific conversion factors used to determine effective dose from dose-length product. Radiology. 2010 Oct;257(1):158-66. doi: 10.1148/radiol.10100047. PMID 20851940
- [Background] van der Molen AJ, Schilham A, Stoop P, Prokop M, Geleijns J. A national survey on radiation dose in CT in The Netherlands. Insights Imaging. 2013 Jun;4(3):383-90. doi: 10.1007/s13244-013-0253-9. Epub 2013 May 15. PMID 23673455
- [Background] Remy-Jardin M, Pistolesi M, Goodman LR, Gefter WB, Gottschalk A, Mayo JR, Sostman HD. Management of suspected acute pulmonary embolism in the era of CT angiography: a statement from the Fleischner Society. Radiology. 2007 Nov;245(2):315-29. doi: 10.1148/radiol.2452070397. Epub 2007 Sep 11. No abstract available. PMID 17848685
- [Background] Lu GM, Zhao Y, Zhang LJ, Schoepf UJ. Dual-energy CT of the lung. AJR Am J Roentgenol. 2012 Nov;199(5 Suppl):S40-53. doi: 10.2214/AJR.12.9112. PMID 23097167
- [Background] Wildberger JE, Klotz E, Ditt H, Mahnken AH, Spuntrup E, Gunther RW. Multi-slice CT for visualization of acute pulmonary embolism: single breath-hold subtraction technique. Rofo. 2005 Jan;177(1):17-23. doi: 10.1055/s-2004-813875. PMID 15657816
- [Background] Mayo J, Thakur Y. Pulmonary CT angiography as first-line imaging for PE: image quality and radiation dose considerations. AJR Am J Roentgenol. 2013 Mar;200(3):522-8. doi: 10.2214/AJR.12.9928. PMID 23436840
- [Background] Pontana F, Faivre JB, Remy-Jardin M, Flohr T, Schmidt B, Tacelli N, Pansini V, Remy J. Lung perfusion with dual-energy multidetector-row CT (MDCT): feasibility for the evaluation of acute pulmonary embolism in 117 consecutive patients. Acad Radiol. 2008 Dec;15(12):1494-504. doi: 10.1016/j.acra.2008.05.018. PMID 19000866
- [Derived] Grob D, Smit E, Prince J, Kist J, Stoger L, Geurts B, Snoeren MM, van Dijk R, Oostveen LJ, Prokop M, Schaefer-Prokop CM, Sechopoulos I, Brink M. Iodine Maps from Subtraction CT or Dual-Energy CT to Detect Pulmonary Emboli with CT Angiography: A Multiple-Observer Study. Radiology. 2019 Jul;292(1):197-205. doi: 10.1148/radiol.2019182666. Epub 2019 May 14. PMID 31084482